CLINICAL TRIAL: NCT04237441
Title: The Results of Pancreatic Operations After the Implementation of Multidisciplinary Team Conference (MDT): A Quality Improvement Study
Brief Title: The Results of Pancreatic Operations After the Implementation of Multidisciplinary Team Conference (MDT):
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, carsten palnaes hansen, chief consultant surgeon, Rigshospitalet, Denmark
Other Study IDs: RH 2015-07, nr. 03616
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDT conference: participants evaluated at MDT conference
  Interventions: Other: number of participants with surgical complications
- no MDT conference: participants not evaluated at MDT conference
  Interventions: Other: number of participants with surgical complications

INTERVENTIONS:
Other: number of participants with surgical complications — observation before and after multidisplinary team conference (MDT) was implemented
  Other Names: number of participants surviving months

SUMMARY:
Background: Centralization has improved the outcome of complex operations including cancer surgery. Moreover, the implementation of multidisciplinary team conferences (MDT) has ameliorated the decision making, but the impact on patient outcome is controversial. The aim of the study was to investigate the outcome of pancreatic surgery in the setting of centralization and upfront multidisciplinary decision making.

DETAILED DESCRIPTION:
Study is a retrospective register study from a prospective database over MDT conferences and patient outcome. End points are quality evaluation regarding postoperative complications and mortality and long-term survival of patients radically operated for pancreatic cancer.

ELIGIBILITY:
Inclusion criteria: all gender seen at multidisciplinary team conference (MDT) Exclusion criteria: all gender not seen at MDT -

-

Ages: 20 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all gender referred to MDT all gender not referred to MDT
Sampling Method: Non-Probability Sample
Enrollment: 7294 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
complications following pancreatic surgery | 14 years
  study from clinical database
survival following pancreatic surgery | 14 years
  study from clinical database

CONTACTS AND LOCATIONS:
Overall Officials: carsten hansen, DMSc, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No